CLINICAL TRIAL: NCT06332157
Title: Postoperative Quality of Recovery After Patients' Undergoing General Anesthesia With Remimazolam Compared to Propofol, A Randomized Non-inferiority Trial
Brief Title: Postoperative Quality of Recovery After General Anesthesia With Remimazolam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-ke-715-1
Record Dates: First submitted 2024-03-17; First posted 2024-03-27 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia Recovery Period

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Anesthesia was induced by pump injection of remimazolam besylate at a rate of 6mg/min. Anesthesia was maintained with 1.0-2.0mg/min remimazolam besylate by continuous pump.
  Interventions: Drug: Remimazolam besylate
- Propofol group (Active Comparator): Anesthesia was induced with propofol injection 2mg/kg intravenously. Anesthesia was maintained by continuous pumping of 6-8mg/kg/h propofol injection.
  Interventions: Drug: Propofol Injection Emulsion

INTERVENTIONS:
Drug: Remimazolam besylate — In Remimazolam group, anesthesia was induced with remimazolam besylate at a rate of 6mg/min and maintained with 1.0-2.0mg/min until the end of surgery.
  Arms: Remimazolam group
Drug: Propofol Injection Emulsion — In Propofol group, anesthesia was induced with propofol injection emulsion at a rate of 2mg/kg and maintained with 6-8mg/kg/h until the end of surgery.
  Arms: Propofol group

SUMMARY:
126 patients undergoing general anesthesia for elective surgery in Beijing Chaoyang Hospital were selected. In the intervention group, anesthesia was induced with remimazolam besylate at a rate of 6mg/min; Anesthesia was maintained with 1.0-2.0mg/min remimazolam besylate by continuous pump. Control group: anesthesia induction, intravenous injection of propofol 2mg/kg; Anesthesia was maintained by continuous pumping of 6-8mg/kg/h propofol. All patients were routinely monitored for vital signs and anesthesia depth after entering the operating room. The patients were followed up after surgery, and the quality of recovery score at 24 hours after surgery was the main study outcome.

DETAILED DESCRIPTION:
This study was a randomized, single-blind, single-center, positive drug controlled, non-inferiority trial. According to the inclusion and exclusion criteria, 126 patients undergoing general anesthesia for elective non-cardiac surgery in Beijing Chaoyang Hospital were selected. In the intervention group, anesthesia was induced with remimazolam besylate at a rate of 6mg/min; Anesthesia was maintained with 1.0-2.0mg/min remimazolam besylate by continuous pump. Control group: anesthesia induction, intravenous injection of propofol 2mg/kg; Anesthesia was maintained by continuous pumping of 6-8mg/kg/h propofol. All patients were routinely monitored for vital signs and anesthesia depth after entering the operating room. After the patient lost consciousness, routine analgesia and muscle relaxants were given, followed by tracheal intubation and mechanical ventilation. During the anesthesia maintenance phase, vital signs and depth of anesthesia were continuously monitored, sedatives and analgesics were continuously pumped, and muscle relaxants were added intermittently as needed. The patients were followed up after surgery, and the quality of recovery score at 24 hours after surgery was the main study outcome.

ELIGIBILITY:
Inclusion Criteria:

1. ASA was classified as I-II
2. The operative time was less than 180 minutes
3. Age ranges from 18 to 65 years
4. Informed consent is signed by all study participants

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with Difficult Airways
3. History of severe neurological and muscular diseases and mental retardation
4. Patients with severe respiratory and circulatory diseases
5. Abnormal liver and kidney function: ALT and/or AST exceeding 2.5 times the upper limit of the medical reference range
6. Urea or urea nitrogen ≥1.5×ULN, serum creatinine greater than the upper limit of normal
7. Take diazole drugs and/or opioids in one month or nearly three months
8. Patients who were allergic to or contraindicated to benzodiazepines, opioids, propofol, flumazenil, naloxone, etc
9. Patients who could not monitor the depth of anesthesia for various reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
15-item quality of recovery scale | 24 hours after surgery
  Patient-measured scales. It was composed of 15 items of five dimensions: physical well-being, physical independence, emotional state, psychological support, and pain. The scale is scored from 0 to 150. Higher scores indicate better quality of recovery.